CLINICAL TRIAL: NCT06062823
Title: An Open-label Phase II Study of EGFR TKI in Patients With Advanced NSCLC Harbouring EGFR Mutations Categorized According to Structural Based Classification
Brief Title: Study of EGFR TKI in Patients With Advanced NSCLC Harbouring EGFR Mutations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS01/02/23
Record Dates: First submitted 2023-08-28; First posted 2023-10-02 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: NSCLC
Keywords: Afatinib; PACC mutation; EGFR mutations
MeSH Terms: interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Afatinib (Experimental): Afatinib given as monotherapy daily in a 28-days cycle.
  Interventions: Drug: Afatinib 40 MG

INTERVENTIONS:
Drug: Afatinib 40 MG — Afatinib 40mg administered orally daily.
  Other Names: Gilotrif

SUMMARY:
The goal of this clinical trial is to explore the efficacy of afatinib in NSCLC harbouring EGFR PACC mutation subtype. The main question it aims to answer is:

Afatinib is active in patients with advanced NSCLC harbouring EGFR PACC mutation subtype.

Participants will undergo screening, follow by treatment if eligible for study participation and then enter follow up phase after study medication has stopped. Patients will take afatinib 40mg daily continuously, until the development of progressive disease or meeting discontinuation criteria. A treatment cycle is defined as 28 days.

DETAILED DESCRIPTION:
This is a multi-center, open-label, phase II study of patients with stage IIIb-IV NSCLC harbouring EGFR PACC mutations.

Before taking the study drug, patients will need to undergo baseline assessments to ensure that they are eligible for the study. Then they will enter treatment period, where afatinib 40mg will be administered daily continuously, until the development of progressive disease or meeting discontinuation criteria. A discontinuation visit will be performed if patients stopped study drug for any reason. Thereafter, patients will be placed on Follow Up visit.

Clinical assessment, routine blood tests and routine imaging:

Physical examinations, imaging, and blood tests will be performed during baseline assessment, on the first day of each treatment cycle, after patients have completed the study and when clinically required by the treating physician. Patients will need to visit the doctor's office approximately 1-2 times every 4 weeks when they are receiving active treatment during the course of the study. More frequent visits may be needed as clinically indicated by the treating physician.

Treatment procedure:

Afatinib will be taken once a day at approximately the same time each day initially starting at a dose of 40mg. Afatinib must be taken on an empty stomach (at least one hour before or at least two hours after a meal).

Research Blood samples:

Blood samples for research will be taken at baseline, before starting cycle 3 and at the time of cancer progression. The estimated total volume of research blood that will be drawn is 10mL (2-3 teaspoons) each time for a total of 30mL.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytologically confirmed NSCLC.
2. No prior systemic therapy for advanced stage disease.
3. Presence of a PACC mutation (detected either in blood or tumour) as defined by Robichaux et al (24). Compound mutations classified as PACC mutations are permitted (24).
4. The presence of measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria (28).
5. Estimated life expectancy of at least 3 months.
6. ECOG performance status 0-1.
7. Age ≥21 years old.
8. Have adequate organ and hematologic function, as defined by:

   * Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤3.0 x upper limit of normal (ULN) or ≤5 times ULN if related to liver metastases.
   * Total serum bilirubin ≤1.5 × ULN (<3.0 × ULN for patients with Gilbert syndrome)
   * Creatinine clearance >=45mL/min (Cockcroft Gault)
   * Absolute neutrophil count ≥1.5 × 10^9/L
   * Platelet count ≥100 × 10^9/L
   * Hemoglobin ≥ 9.0 g/dL
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
10. For female patients of childbearing potential, have a negative pregnancy test documented ≤ 14 days prior to start of study medication.
11. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use a highly effective form of contraception with their sexual partners during the dosing period and for a period of at least 4 months after the end of treatment. Evidence of non-child-bearing potential is fulfilled by one of the following criteria at screening:

    * The post-menopausal period defined as age ≥50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
    * Women <50 years old they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range.
    * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not a tubal ligation
12. Signed written informed consent.

Exclusion Criteria:

1. Prior EGFR TKI therapy.
2. Prior chemotherapy for Stage IIIB/IV adenocarcinoma of the lung. Neo-/adjuvant chemotherapy, CT-RT or RT is permitted if it has been elapsed for ≥12 months prior to disease progression.
3. Have been diagnosed with another primary malignancy other than NSCLC, except for adequately treated non melanoma skin cancer or cervical cancer in situ; definitively treated non metastatic prostate cancer; or patients with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
4. Known leptomeningeal carcinomatosis.
5. Unstable spinal cord compression/brain metastases unless asymptomatic and not requiring steroids for at least 2 weeks prior to the start of study treatment. For patients with brain metastases, gamma knife or stereotactic brain surgery is allowed prior to study treatment.
6. Symptomatic and untreated spinal cord compression.
7. Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to: myocardial infarction within 6 months prior to study enrolment; unstable angina within 6 months prior to study enrolment; congestive heart failure within 6 months prior to study enrolment; history of clinically significant atrial arrhythmia (including clinically significant bradyarrhythmia), as determined by the treating physician; any history of clinically significant ventricular arrhythmia; prolonged QTc.
8. Had a cerebrovascular accident or transient ischemic attack within 6 months prior to enrolment.
9. Major surgery within 4 weeks of starting study treatment and patients must have recovered from any effects of any major surgery. Minor surgery is allowed.
10. Radiotherapy to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks before the study entry.
11. Inability to swallow oral medication.
12. Refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection that would preclude adequate absorption of afatinib.
13. Have a history or the presence at baseline of pulmonary interstitial disease, drug-related pneumonitis, or radiation pneumonitis.
14. Have an ongoing or active infection, including, but not limited to, the requirement for intravenous antibiotics.
15. Have a known history of human immunodeficiency virus infection or active hepatitis B or C infection, active tuberculosis.
16. Have a known or suspected hypersensitivity to afatinib or its excipients.
17. Are pregnant, planning a pregnancy, or breastfeeding.
18. Males and females of reproductive potential who are not using an effective method of contraception and females who are pregnant or breastfeeding or have a positive serum pregnancy test prior to study entry.
19. Previous allogeneic bone marrow transplant.
20. Have any condition or illness that, in the opinion of the investigator, would compromise patient safety or interfere with the study treatment.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | At baseline and every 8 weeks for the first 6 cycles, every 12 weeks from cycle 7 to 12 and every 16 weeks from cycle 13 onwards (each cycle is 28 days)
  Defined as best overall response (Complete Response or Partial Response) across all assessment time-points according to RECIST criteria v1.1

SECONDARY OUTCOMES:
Progression free survival | within 4 weeks from starting treatment and every 8 weeks for the first 6 cycles, every 12 weeks from cycle 7 to 12 and every 16 weeks from cycle 13 onwards (each cycle is 28 days)
  Defined as the time from the date of study enrolment to the first date of documented disease progression
Overall survival | 48 months
  Defined as the time from the date of randomisation until documented progression (according to RECIST v1.1) or death
Duration of response | every 8 weeks for the first 6 cycles, every 12 weeks from cycle 7 to 12 and every 16 weeks from cycle 13 onwards (each cycle is 28 days)
  Defined as the time from first documented Complete Response or Partial Response to the time of radiological progression or death, whichever occurs earlier.
Time to treatment failure | 48 months
  Defined as the time from afatinib treatment to the time of treatment discontinuation for any reason including disease progression, treatment toxicity, and death
Number of participant with treatment related toxicities | 48 months
  Toxicities will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) toxicity grading Version 5

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Sooi, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonomi PD. Implications of key trials in advanced nonsmall cell lung cancer. Cancer. 2010 Mar 1;116(5):1155-64. doi: 10.1002/cncr.24815. PMID 20087963
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Planchard D, Smit EF, Groen HJM, Mazieres J, Besse B, Helland A, Giannone V, D'Amelio AM Jr, Zhang P, Mookerjee B, Johnson BE. Dabrafenib plus trametinib in patients with previously untreated BRAFV600E-mutant metastatic non-small-cell lung cancer: an open-label, phase 2 trial. Lancet Oncol. 2017 Oct;18(10):1307-1316. doi: 10.1016/S1470-2045(17)30679-4. Epub 2017 Sep 11. PMID 28919011
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Shaw AT, Ou SH, Bang YJ, Camidge DR, Solomon BJ, Salgia R, Riely GJ, Varella-Garcia M, Shapiro GI, Costa DB, Doebele RC, Le LP, Zheng Z, Tan W, Stephenson P, Shreeve SM, Tye LM, Christensen JG, Wilner KD, Clark JW, Iafrate AJ. Crizotinib in ROS1-rearranged non-small-cell lung cancer. N Engl J Med. 2014 Nov 20;371(21):1963-71. doi: 10.1056/NEJMoa1406766. Epub 2014 Sep 27. PMID 25264305
- [Background] Solomon BJ, Mok T, Kim DW, Wu YL, Nakagawa K, Mekhail T, Felip E, Cappuzzo F, Paolini J, Usari T, Iyer S, Reisman A, Wilner KD, Tursi J, Blackhall F; PROFILE 1014 Investigators. First-line crizotinib versus chemotherapy in ALK-positive lung cancer. N Engl J Med. 2014 Dec 4;371(23):2167-77. doi: 10.1056/NEJMoa1408440. PMID 25470694
- [Background] Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, Dechaphunkul A, Imamura F, Nogami N, Kurata T, Okamoto I, Zhou C, Cho BC, Cheng Y, Cho EK, Voon PJ, Planchard D, Su WC, Gray JE, Lee SM, Hodge R, Marotti M, Rukazenkov Y, Ramalingam SS; FLAURA Investigators. Osimertinib in Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Jan 11;378(2):113-125. doi: 10.1056/NEJMoa1713137. Epub 2017 Nov 18. PMID 29151359
- [Background] Planchard D, Popat S, Kerr K, Novello S, Smit EF, Faivre-Finn C, Mok TS, Reck M, Van Schil PE, Hellmann MD, Peters S; ESMO Guidelines Committee. Metastatic non-small cell lung cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv192-iv237. doi: 10.1093/annonc/mdy275. No abstract available. PMID 30285222
- [Background] Lynch TJ Jr, Kim ES, Eaby B, Garey J, West DP, Lacouture ME. Epidermal growth factor receptor inhibitor-associated cutaneous toxicities: an evolving paradigm in clinical management. Oncologist. 2007 May;12(5):610-21. doi: 10.1634/theoncologist.12-5-610. PMID 17522250
- [Background] Lacouture ME, Schadendorf D, Chu CY, Uttenreuther-Fischer M, Stammberger U, O'Brien D, Hauschild A. Dermatologic adverse events associated with afatinib: an oral ErbB family blocker. Expert Rev Anticancer Ther. 2013 Jun;13(6):721-8. doi: 10.1586/era.13.30. Epub 2013 Mar 18. PMID 23506519
- [Background] Aw DC, Tan EH, Chin TM, Lim HL, Lee HY, Soo RA. Management of epidermal growth factor receptor tyrosine kinase inhibitor-related cutaneous and gastrointestinal toxicities. Asia Pac J Clin Oncol. 2018 Feb;14(1):23-31. doi: 10.1111/ajco.12687. Epub 2017 May 2. PMID 28464435
- [Background] Yang JC, Sequist LV, Geater SL, Tsai CM, Mok TS, Schuler M, Yamamoto N, Yu CJ, Ou SH, Zhou C, Massey D, Zazulina V, Wu YL. Clinical activity of afatinib in patients with advanced non-small-cell lung cancer harbouring uncommon EGFR mutations: a combined post-hoc analysis of LUX-Lung 2, LUX-Lung 3, and LUX-Lung 6. Lancet Oncol. 2015 Jul;16(7):830-8. doi: 10.1016/S1470-2045(15)00026-1. Epub 2015 Jun 4. PMID 26051236
- [Background] Robichaux JP, Le X, Vijayan RSK, Hicks JK, Heeke S, Elamin YY, Lin HY, Udagawa H, Skoulidis F, Tran H, Varghese S, He J, Zhang F, Nilsson MB, Hu L, Poteete A, Rinsurongkawong W, Zhang X, Ren C, Liu X, Hong L, Zhang J, Diao L, Madison R, Schrock AB, Saam J, Raymond V, Fang B, Wang J, Ha MJ, Cross JB, Gray JE, Heymach JV. Structure-based classification predicts drug response in EGFR-mutant NSCLC. Nature. 2021 Sep;597(7878):732-737. doi: 10.1038/s41586-021-03898-1. Epub 2021 Sep 15. PMID 34526717
- [Background] Russo A, Franchina T, Ricciardi G, Battaglia A, Picciotto M, Adamo V. Heterogeneous Responses to Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitors (TKIs) in Patients with Uncommon EGFR Mutations: New Insights and Future Perspectives in this Complex Clinical Scenario. Int J Mol Sci. 2019 Mar 21;20(6):1431. doi: 10.3390/ijms20061431. PMID 30901844
- [Background] Kobayashi Y, Mitsudomi T. Not all epidermal growth factor receptor mutations in lung cancer are created equal: Perspectives for individualized treatment strategy. Cancer Sci. 2016 Sep;107(9):1179-86. doi: 10.1111/cas.12996. Epub 2016 Aug 9. PMID 27323238
- [Background] Gu L, Huang H, Xu Z, Niu X, Li Z, Xia L, Yu Y, Lu S. Landscape and Predictive Significance of the Structural Classification of EGFR Mutations in Chinese NSCLCs: A Real-World Study. J Clin Med. 2022 Dec 28;12(1):236. doi: 10.3390/jcm12010236. PMID 36615035
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835